CLINICAL TRIAL: NCT01814501
Title: A Phase II Study of Panitumumab in Combination With FOLFIRI After Progression on FOLFIRI Plus Bevacizumab in KRAS(Kirsten Rat Sarcoma) and NRAS Wild-Type Metastatic Colorectal Cancer.
Brief Title: Panitumumab and Chemotherapy in Patients With Advanced Colorectal Cancer After Prior Therapy With Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Hays (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, John Hays, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-11131; NCI-2013-00432 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-25; First posted 2013-03-20 (Estimated); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IV Colon Cancer; Stage IV Rectal Cancer
Keywords: Metastatic colon cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Panitumumab; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (panitumumab, combination chemotherapy) (Experimental): 5-Fluorouracil, irinotecan, and panitumumab
  Interventions: Biological: panitumumab; Drug: irinotecan hydrochloride; Drug: fluorouracil; Drug: leucovorin calcium

INTERVENTIONS:
Biological: panitumumab — Each vial of panitumumab will contain 20 mL of a sterile protein solution containing a 20-mg/mL solution of panitumumab. The vial will contain approximately 400mg of panitumumab and is for single dose use only.
  Other Names: ABX-EGF; MOAB ABX-EGF; monoclonal antibody ABX-EGF; Vectibix
Drug: irinotecan hydrochloride — Diluted with 5% dextrose (D5W) to a total volume of 500 mL and infused intravenously over 90 minutes. Nothing else should be added to the bag. Patients will be given a dose of 180 mg/M2 by intravenous infusion.
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: fluorouracil — Administered intravenously. A bolus of 400 mg/m2 to be followed by a continuous infusion over 46 hrs at a dose of 2400mg/m2.
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: leucovorin calcium — Leucovorin will be administered at a dose of 200 mg/m2 over 120 minutes prior to the 5-FU bolus. Leucovorin may be run simultaneously with irinotecan infusion via y-site connection.
  Other Names: CF; CFR; LV

SUMMARY:
This phase II trial studies how well panitumumab and combination chemotherapy works in treating patients with metastatic colorectal cancer previously treated with combination chemotherapy and bevacizumab. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving panitumumab and combination chemotherapy together may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the median progression-free survival in patients treated with leucovorin calcium, fluorouracil, and irinotecan hydrochloride (FOLFIRI) and panitumumab for K-ras and NRAS wild-type, metastatic colorectal carcinoma who have already progressed on FOLFIRI + Bevacizumab.

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of toxicities of the regimens. II. To determine overall response rate. III. To determine the median overall survival and the overall survival rate at 1 year.

OUTLINE:

Patients receive panitumumab intravenously (IV) over 60-90 minutes, leucovorin calcium IV over 90 minutes, fluorouracil IV continuously over 46 hours, and irinotecan hydrochloride IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced adenocarcinoma of the colon or rectum not curable with surgery or radiotherapy and have been previously treated for their disease with FOLFIRI plus bevacizumab in the first line metastatic setting; patients will only be eligible if their last line of therapy prior to enrolling onto the study was FOLFIRI and bevacizumab received no more than 6 months prior to enrolling in this study; they should have been treated with FOLFIRI plus bevacizumab until disease progression is radiographically documented
* Patients' tumors will need to tested for the K-RAS and N-RAS mutation status; only those patients with wild-type or unmutated K-RAS and N-RAS oncogene are eligible to participate in this study
* Provide written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* Prior cetuximab is allowed in the adjuvant but not in the metastatic setting, but must have been completed at least 6 months before starting this trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy greater than 12 weeks
* No active brain metastasis; previously surgically treated or irradiated lesions are allowed if not clinically active
* Has a negative serum pregnancy test within 7 days prior to registration (female patients of childbearing potential)
* Ability to understand and willingness to sign a written informed consent
* No history of severe reactions to fluorouracil (5-FU), irinotecan (irinotecan hydrochloride), or a monoclonal antibody
* Leukocytes >= 3000/uL
* Absolute neutrophil count >= 1500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 mg/dL
* Total bilirubin =< 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 X ULN (or < 5 x ULN with liver metastases)
* Creatinine clearance (CrCl) >= 30 ml/min (Cockroft-Gault equation)
* Magnesium >= lower limit of normal
* Measurable disease is required according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* The effects of Panitumumab on the developing human fetus are unknown; for this reason and because monoclonal antibodies as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and up to 6 months after completing therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Pregnant or lactating women; women of childbearing potential with either a positive or no pregnancy test at baseline; woman or men of childbearing potential not using a reliable and appropriate contraceptive method; (postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential)
* Sexually active males unwilling to practice contraception during the study and 6 months beyond
* Uncontrolled intercurrent illness including but not limited to clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction within the last 12 months, and serious concurrent infections
* History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest computed tomography (CT) scan
* KRAS or NRAS mutant tumors
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as >= Common Toxicity Criteria [CTC] grade 2 [Common Terminology Criteria for Adverse Events (CTCAE) version 4.0])
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) =< 1 year
* Bevacizumab within the last 4 weeks before starting treatment on trial
* Patient is more than 6 months since the last dose of FOLFIRI
* Patients who have required toxicity related dose reductions of no less than 50% of the original dose of infusional 5-FU and/or irinotecan during the administration of FOLFIRI + bevacizumab
* Prior exposure to panitumumab in any setting
* Prior exposure to cetuximab in the metastatic (stage IV) setting
* Radiotherapy =< 14 days prior to enrollment; patients must have recovered from all radiotherapy-related toxicities
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil, leucovorin (leucovorin calcium), irinotecan, or panitumumab
* Treatment for other carcinomas within the last three years, except cured non-melanoma skin and treated in-situ cervical cancer
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation
* Major surgery within 4 weeks of the start of study treatment, without complete recovery
* Unwillingness to give written informed consent
* Unwillingness to participate or inability to comply with the protocol for the duration of the study
* Patients with human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS) and those severely immunocompromised will be excluded; however, no patients will be tested for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hays, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Panitumumab, Combination Chemotherapy): 5-Fluorouracil, irinotecan, and panitumumab
  panitumumab: Given IV
  irinotecan hydrochloride: Given IV
  fluorouracil: Given IV
  leucovorin calcium: Given IV
Period: Overall Study
Arm/Group | Treatment (Panitumumab, Combination Chemotherapy)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Panitumumab, Combination Chemotherapy)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Continuous variables will be expressed by means, standard deviations and 95% confidence intervals. Estimated using the Kaplan-Meier estimator with confidence interval calculated based on the Brookmeyer-Crowley method.
Time Frame: Time from study day 1 to the time the patient is first recorded as having disease progression or death, assessed up to 3 years
Measure: Mean (95% Confidence Interval); unit: days to progression
Arm/Group | Treatment (Panitumumab, Combination Chemotherapy)
Number analyzed (Participants) | 16
days to progression | 255.921 [189.162 to 322.680]

2. Secondary Outcome: Frequency and Severity of Toxicities of the Regimens, Graded According to the NCI CTCAE v4.0
Description: Frequencies will be computed for discrete data. Toxicities graded per NCI CTCAE v4.0 grade 3, 4, 5
Time Frame: Up to 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Panitumumab, Combination Chemotherapy)
Number analyzed (Participants) | 16
percentage of patients
  Increased ALT | 6.3
  Increased AST | 6.3
  Diarrhea | 6.3
  Fatigue | 12.5
  Gastrointestional disorders | 6.3
  Hypertension | 12.5
  Hypokalemia | 6.3
  Hypomagnesemia | 12.5
  Hyponatremia | 12.5
  Lymphocyte count decreased | 12.5
  Lymphocyte count increased | 6.3
  Mucositis oral | 25
  Neoplasms benign, malignant and unspecified | 6.3
  Neutrophil count decreased | 6.3
  Palmar-plantar erythrodysesthesia syndrome | 6.3
  Pruritus | 6.3
  Skin and subcutaneous tissue disorders | 6.3
  Sleep apnea | 6.3
  White blood cell decreased | 6.3

3. Secondary Outcome: Proportion of Participants With Overall Response Rate, as Described in RECIST v1.1 Criteria
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Panitumumab, Combination Chemotherapy)
Number analyzed (Participants) | 16
proportion of participants | 0.1875 [0.0405 to 0.4565]

4. Secondary Outcome: Overall Survival
Description: Continuous variables will be expressed by means, standard deviations and 95% confidence intervals. Kaplan-Meier estimator will be used.
Time Frame: Time from study day 1 to the date of death or the last date the patient was known to be alive, assessed up to 3 years
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Treatment (Panitumumab, Combination Chemotherapy)
Number analyzed (Participants) | 16
days | 471 [32.340 to 909.660]

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from baseline to study follow-up using the National Cancer Institute (NCI) CTCAE version 4.0, an average of 4 years.
Arm/Group | Treatment (Panitumumab, Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 15/16
Serious Adverse Events (participants affected / at risk) | 16/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Panitumumab, Combination Chemotherapy) (N=16)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Lymphocyte count increased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Panitumumab, Combination Chemotherapy) (N=16)
Abdominal Pain (Gastrointestinal disorders) | 8 (8)
Activated partial thromboplastin time prolonged (Investigations) | 5 (5)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 5 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 13 (13)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Dizziness (Nervous system disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 8 (8)
Eye disorders - Other, specify (Eye disorders) | 3 (3)
Eye pain (Eye disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Headache (Nervous system disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (13)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Infusion related reaction (Immune system disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Localized edema (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (8)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (9)
Neutrophil count decreased (Investigations) | 4 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Paronychia (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Platelet count decreased (Investigations) | 4 (4)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7 (7)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT01814501/Prot_SAP_000.pdf